CLINICAL TRIAL: NCT05431842
Title: Analysis of Reliability and Validity of Urdu Version of Functional Gait Assessment Scale Among Pakistani Geriatric Population
Brief Title: Urdu Version of Functional Gait Assessment Scale: Reliability and Validity Study
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00265
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Stroke
Keywords: Functional Gait Assessment Scale; Urdu Version; Reliability; Validity; Stroke; Geriatric Population
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of study is to translate and culturally adapt Functional Gait Assessment Scale into Urdu language and to investigate the reliability and validity in Pakistani Stroke patients. Also check its correlation with Berg Balance Scale and Barthel Index

DETAILED DESCRIPTION:
The English version of the Functional Gait Assessment Scale will be translated and culturally adapted as per previous recommendation. In geriatric population, Urdu Version of Functional Gait Assessment Scale will distributed among 160 participants choose by convenience sampling technique based on pre-defined inclusion and exclusion criteria.To test inter and intra-observer reliability of the final Urdu Version of Functional Gait Assessment Scale, Barthel Index and Berg Balance Scale, questionnaire will be filled on the same day. Data will be entered and analyzed using Statistical Package of Social Sciences Version 24. Internal consistency will be analyzed with Cronbach alpha value. Test- retest reliability will be assessed for intra-class correlation coefficient. The Urdu Version of Functional Gait Assessment Scale was evaluated for content validity, construct validity, criterion validity and responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years
* Post stroke patients past 3 months
* Both gender patients are included

Exclusion Criteria:

* Patient suffering from any neurological disorder
* Patient suffering from any musculoskeletal disorder
* Patients who are post stroke less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pakistani population post-stroke over the age of 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Functional Gait Assessment Scale | 1st day
  Functional Gait Assessment Scale is used to evaluate the constructions of balance and gait in ambulatory stroke patients. Number of Test Items: 10 Scoring: Each item is scored on an ordinal scale from 0 - 3, with 0 = severe impairment, 1 = moderate impairment, 2 = mild impairment, 3 = normal ambulation, Thus, the highest score is 30/30.
Barthel Index | 1st day
  Barthel Index is use to assess the level of independence and autonomy of stroke patient in performing ADLs. It is a list of 10 elementary ADLs: feeding, grooming, bathing, dressing, bowel and bladder care, toilet use, ambulation, transfers, and stair climbing. The activities are rated through time taken and assistance used by patient. Score ranges from 0-100.
Berg Balance Scale | 1st day
  the berg balance scale is an objective assessment of balance performance based on 14 items common to daily activities. it is a 14 items scale that rate 0 (unable to perform) to 4 (normal performance) for each item. the total score is 56 points, high score higher balance ability

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No